CLINICAL TRIAL: NCT03267745
Title: Effects of Amino Acid Formulation on Healthy Men Undergoing Unilateral Knee Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Axcella Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3365
Record Dates: First submitted 2017-08-09; First posted 2017-08-30 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Muscle Atrophy
Keywords: protein; skeletal muscle; immobilization
MeSH Terms: conditions — Muscular Atrophy | interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: 2 groups of 10 each will be randomized to receive amino acid supplementation or placebo for 28 days during which they will have one leg immobilized by a removable brace.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sachets with the supplement will be blinded to the participant, and research assistants. Outcomes assessors will be blinded to condition as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino Acid (Experimental): Subjects in this arm will receive amino acid supplementation (23.7g) 3 times daily for 28 days. Amino acids will be provided in powder form to be dissolved in 8oz of water. Participants will also undergo single-leg immobilization (Breg brace) for 7 days (days 8-15) during the 28 day study period.
  Interventions: Dietary Supplement: Amino Acid; Device: Breg Brace single-leg immobilization
- Placebo (Placebo Comparator): Subjects in this arm will receive placebo 3 times daily for 28 days. Placebo will consist of 23.7g of excipient-matched placebo in water. Participants will also undergo single-leg immobilization (Breg brace) for 7 days (days 8-15) during the 28 day study period.
  Interventions: Device: Breg Brace single-leg immobilization; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Amino Acid — 23.7 g amino acid 3 times daily for 28 days
  Arms: Amino Acid
Device: Breg Brace single-leg immobilization — 7 days of single leg immobilization; randomized to leg; knee brace will be worn in a fixed flexion position at 140°.
  Other Names: Breg brace
Other: Placebo — Excipient-matched placebo 3 times daily for 28 days
  Arms: Placebo

SUMMARY:
This is a safety and tolerability study investigating the effect of an amino acid formulation in healthy volunteers during and after limb immobilization.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy, non-smoking
2. Willing and able to provide informed consent
3. Men age 20-45 years
4. BMI between 25 and 35 kg/m2

Exclusion Criteria:

1. Smoker;
2. Subject has any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements;
3. History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years;
4. Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder (requiring ongoing medical care), or metabolic/endocrine disorder (e.g., diabetes, high cholesterol, elevated fasting blood sugar) or other disease that would preclude oral protein supplement ingestion and/or assessment of safety and study objectives;
5. Any cachexia-related condition (e.g., relating to cancer, tuberculosis or human immunodeficiency virus infection and acquired immune deficiency syndrome) or any genetic muscle diseases or disorders;
6. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing);
7. Subject participated in a study of an investigational product less than 60 days or 5 half-lives of the investigational product, whichever is longer, before enrollment in this study;
8. Hypersensitivity to any of the components of the test product;
9. Excessive alcohol consumption (>21 units/week); (> 21 standard drinks/wk); e.g., 18oz glass of 5% beer - 1.5 standard drinks, a 750 mL bottle of 12% wine = 5 standard drinks.
10. Known sensitivity or allergy to amino acids or any ingredient in the test formulations;
11. Prior gastrointestinal bypass surgery (Lapband, etc.), irritable bowel disease or irritable bowel syndrome;
12. History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy (up to 81mg of baby aspirin per day taken as a prophylactic is permitted);
13. Personal or family history of clotting disorder or deep vein thrombosis. Deep vein thrombosis is a serious, and potentially lethal, medical condition, therefore, it is imperative if you have personal or family history it is disclosed this to the research staff.
14. Concomitant use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), any anabolic steroid, creatine, whey protein supplements, casein or branched-chain amino acids (BCAAs) within 45 days prior to Screening;
15. Contraindications to an MRI scan (e.g. subjects with non-removable ferromagnetic implants, pacemakers, aneurysm clips or other foreign bodies, or subjects with claustrophobic symptoms that would contraindicate an MRI scan).
16. Hemoglobin <11.5mg/dl at Screening;
17. Platelets <150,000/uL (150x109/L) at Screening.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in muscle atrophy | day 0, day 8, day 15 and day 28
  To determine the impact of an amino acid formulation on muscle atrophy after 7 days of amino acid supplementation followed by 7 days of single leg immobilization and 14 days of recovery post-immobilization muscle atrophy will be assessed utilizing percutaneous muscle biopsy to quantify fibre size in the vastus lateralis.

SECONDARY OUTCOMES:
Change in muscle strength | day 0, day 8, day 15 and day 28
  Strength will be measured using a Biodex.
Change in muscle size | day 0, day 8, day 15 and day 28
  Muscle size will be assessed via MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holloway TM, McGlory C, McKellar S, Morgan A, Hamill M, Afeyan R, Comb W, Confer S, Zhao P, Hinton M, Kubassova O, Chakravarthy MV, Phillips SM. A Novel Amino Acid Composition Ameliorates Short-Term Muscle Disuse Atrophy in Healthy Young Men. Front Nutr. 2019 Jul 10;6:105. doi: 10.3389/fnut.2019.00105. eCollection 2019. PMID 31355205